CLINICAL TRIAL: NCT05602779
Title: Leveraging Noninvasive Transcutaneous Vagus Nerve Stimulation and Smartphone Technology to Reduce Suicidal Behaviors and Suicide Among Highly Vulnerable Adolescents
Brief Title: Leverage Noninvasive Transcutaneous Vagus Nerve Stimulation to Reduce Suicidal Behaviors in Vulnerable Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: University of Rochester (Other); University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Kristin Valentino, Professor of Psychology, University of Notre Dame
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-08-7372
Record Dates: First submitted 2022-10-06; First posted 2022-11-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Self Harm; Suicidal Ideation
Keywords: Self Harm; Suicide Prevention
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: There will be four distinct treatment groups, each participant will be randomly assigned to one of the four groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- tVNS Program + Control app (Experimental): Adolescents will self-administer 30-minute tVNS (i.e., nerve stimulation) sessions daily for 30 days. They will receive a daily text message on their phone to remind them about their session. They will have access to MindTiles where they will complete daily puzzles on their own. In addition, they will answer a 2-3 minute self-report survey on their current thoughts, feelings, and behaviors once a day for 30 days. They will receive a text message with a link to Qualtrics, a secure online platform where they will complete the survey.
  Interventions: Device: tVNS Program
- Phone App Program + Sham tVNS (Experimental): Adolescents will use a specially designed phone app (MindTiles) to communicate with peer to help them cope with emotions, and to foster connection with peers to establish social connections. In addition, they will answer a 2-3 minute self-report survey on their current thoughts, feelings, and behaviors once a day for 30 days. They will receive a text message with a link to Qualtrics, a secure online platform where they will complete the survey. Adolescents will also self-administer 30-minute sham tVNS (i.e., nerve stimulation) sessions daily for 30 days; these sessions will include no actual stimulation.
  Interventions: Other: Phone App Program
- tVNS and Phone App Program (Experimental): Adolescents will self-administer 30-minute tVNS (i.e., nerve stimulation) sessions daily for 30 days. Adolescents will also use a specially designed phone app (MindTiles) to communicate with a peer to help them cope with emotions, and to foster connection with peers to establish social connections. They will receive a daily text message on their phone to remind them about their session. In addition, they will answer a 2-3 minute self-report survey on their current thoughts, feelings, and behaviors once a day for 30 days. They will receive a text message with a link to Qualtrics, a secure online platform where they will complete the survey.
  Interventions: Combination Product: tVNS and Phone App Program
- Sham tVNS + Control App (Sham Comparator): Adolescents will self-administer 30-minute sham tVNS (i.e., nerve stimulation) sessions daily for 30 days; these sessions will include no actual stimulation.They will receive a daily text message on their phone to remind them about their session. They will also have access to MindTiles where they will complete daily puzzles on their own. They will answer a 2-3 minute self-report survey on their current thoughts, feelings, and behaviors once a day for 30 days. They will receive a text message with a link to Qualtrics, a secure online platform where they will complete the survey.
  Interventions: Other: Sham tNVS and Control App

INTERVENTIONS:
Device: tVNS Program — Participants will use the Neuvana Xen device 30 minutes a day for 30 days. The device delivers stimulation through the left ear via an ear bud. Participants can use the device at any time of day.
  Arms: tVNS Program + Control app
Other: Phone App Program — Participants will have access to a specially designed phone app (MindTiles) in order to play a game designed for this study. Participants in the active intervention will be able to connect with a fellow participant who is matched as their peer for social support and they will complete a daily puzzle together and respond to a conversational prompt to encourage communication.
  Arms: Phone App Program + Sham tVNS
Combination Product: tVNS and Phone App Program — Participants will have both the Neuvana Xen Device and the full version of our program's phone app. They will use the device and full app access for 30 days.
  Arms: tVNS and Phone App Program
Other: Sham tNVS and Control App — Participants will have access to our program's phone app so the can complete the daily puzzle on their own. They will also engage in a sham tVNS session for 30min per day for 30 days during which no stimulation is provided.
  Arms: Sham tVNS + Control App

SUMMARY:
Suicidal thoughts, suicide attempts, and suicide are increasingly common in adolescence.

Current face-to-face prevention approaches are of limited effectiveness, rely on extensive resources, and are at odds with adolescents' digital preferences. We will evaluate two unconventional but promising interventions delivered to 13- to 17-year-olds: transcutaneous vagus nerve stimulation to target emotion dysregulation, and a peer-support smartphone app to combat social isolation. If effective, these digitally-delivered interventions could reach far more adolescents at far lower cost than current approaches.

DETAILED DESCRIPTION:
Over the past two decades, suicide rates have increased nearly 35% in the U.S., with upward trends in nearly all demographic groups. Further increases have occurred since the COVID-19 pandemic began. Despite ambitious goals for reducing suicides and significant federal and private investment, suicide rates continue to rise unabated. To date, the predominant approach to mitigating suicide risk in the U.S. is secondary prevention. Typically, these programs identify risk of recurrence among those who have already attempted suicide at least once. Although secondary prevention is crucial, the majority of deaths by suicide occur on first attempt. Thus, targeted primary prevention earlier in development is essential. Most current primary prevention programs are intensive, expensive, and delivered by highly trained mental health providers, who are in short supply. Traditional face-to-face therapy is also unavailable to many who live in underserved communities, and disliked by adolescents, who much prefer digital delivery on their devices. This high-risk, high-reward proposal addresses these limitations and needs. We use an experimental therapeutics approach to evaluate the independent and combined efficacies of two unconventional but scalable interventions: transcutaneous vagus nerve stimulation (tVNS) to target emotion dysregulation, and a peer-support smartphone app to combat social isolation. These low-cost interventions, which hold strong promise but have not been used before, can reach large numbers of adolescents, with much potential to reduce prospective suicide risk. We will enroll 212 adolescents, ages 13-17 years, who show elevations on at least two prominent risk factors for suicide (e.g., self-injury, maltreatment).

Using a 2 × 2 design, adolescents will be assigned randomly to receive 30 days of treatment with:

1. tVNS to target emotion dysregulation,
2. a peer-support phone app to target social isolation,
3. tVNS + a peer-support phone app, or
4. enhanced treatment as usual with monitoring and access to resources.

Intervention effects on mechanisms (emotion dysregulation, social isolation) proximal efficacy signals (e.g., physiological reactivity, self-harm) and target outcomes (suicidal ideation, suicidal behaviors) will be evaluated immediately post-intervention and at one-year follow-up. Treatment data will be monitored daily to fine-tune dosing of both interventions. This transformative and innovative proposal tests two novel, scalable preventive interventions designed to "meet adolescents where they are" by using digital technologies to address core mechanisms of suicide risk.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 13 and 17 years,
* Daily access to a smartphone
* Attend in person meetings in South Bend, IN or Rochester, NY. and,

Two of the following which will be scored during the phone screen:

* High scores on social isolation
* High scores on emotion dysregulation
* Has engaged in NSSI (inclusive of a single act)
* High T-scores on impulsivity,
* High T-scores on depression
* Engages in alcohol or other substance use

Exclusion Criteria:

* Parent reported autism or schizophrenia
* Implanted pacemaker or cardiac defibrillator, other implanted or metallic device
* Pregnant or breast feeding
* History of seizures or epilepsy
* TMJ Disorder
* Bells' Palsy
* Impaired cranial nerve function
* Facial Pain

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline to Follow-up Assessments in Self-Injurious Thoughts and Behaviors over one year | 30 Days; One Year
  Teens will be assessed at baseline visits for self-injurious thoughts and behaviors (non-suicidal self-injury (NSSI), suicidal ideation (SI), suicide attempts (SA)). They will complete measures individually on the Qualtrics Survey (SIQ) as well as participate in a face-to-face interview with a trained staff member to assess their level of NSSI, SI, and SA (CSSRS, DSHI).
  All participants will repeat these tasks at all visits (post-treatment, one-year follow-up). We expect teens who have used the active tVNS device will show improved responses (e.g., decreases in NSSI and SI). Teens who have engaged in the peer-matched MindTiles condition will show improved responses in SI, SA, and NSSI. For both conditions we will examine rates of self-injurious thoughts and behaviors in the treatment arms in relation to national norms. We plan to examine between group change across treatment groups as well as within-person change at 30 days and one year post intervention.

SECONDARY OUTCOMES:
Change from Baseline to Follow-up Assessments in Emotion Dysregulation | 30 Days; One Year
  Some teens will be randomized to the active tVNS condition where they will receive daily stimulation to their vagus nerve, which should modulate emotion dysregulation. Each participating teen will complete questionnaires regarding emotion dysregulation on the Qualtrics survey (Difficulties in Emotion Regulation Scale (DERS)) at all timepoints. We anticipate those who are randomized to the active tVNS condition will show improvement in emotion dysregulation at 30 days and one year post treatment relative to the other treatment arms, as well as show improved within-person change.
Change from Baseline to Follow-up Assessments in Social Connection and Loneliness | 30 Days; One Year
  Some teens will be assigned to using the peer support phone app where they will be matched with another teen in the study. They will play a cooperative game with each other, and be able to text and share thoughts, feelings, etc. with each other during the 30 days intervention period. The peer-matched MindTiles app is expected to improve teen's self-reported feelings of isolation and loneliness.
  Each participating teen will complete questions regarding feelings of loneliness and social isolation on the Qualtrics survey during all lab visits. We are using the 3 Item UCLA Loneliness scale and the INQ-15. We plan to examine between group change across treatment groups as well as within-person change at 30 days and one year post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Valentino, PhD, Principal Investigator — University of Notre Dame
Locations (2):
- United States (2):
  - University of Notre Dame, South Bend, Indiana
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data outside of the study team.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT05602779/SAP_000.pdf